CLINICAL TRIAL: NCT02415686
Title: Cardiac Arrhythmias in Dravet Syndrome: an Observational, International, Multicentre Study
Brief Title: Cardiac Arrhythmias in Dravet Syndrome
Status: Completed | Type: Observational
Sponsor: Stichting Epilepsie Instellingen Nederland (Other)
Collaborators: Epilepsiefonds (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL48765.058.15
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
Keywords: Dravet syndrome; Sudden Unexpected Death in Epilepsy (SUDEP); Arrhythmias
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Sudden Unexpected Death in Epilepsy; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
SUMMARY

Rationale:

People with Dravet Syndrome (DS), a rare epilepsy syndrome, have a high risk of Sudden Unexpected Death in Epilepsy (SUDEP). Mouse models indicated that the responsible sodium channel mutation (SCN1A) not only alters cortical excitability but also increases the propensity to arrhythmias. Little is known yet about the prevalence of seizure-induced arrhythmias in human DS subjects.

Objective:

To assess the prevalence of cardiac arrhythmias in DS and to compare the prevalence of cardiac arrhythmias between DS subjects and subjects with other types of epilepsy.

Study design:

Observational study.

Study population:

Subjects with Dravet syndrome and a known pathogenic SCN1A mutation, seizure frequency ≥ 1/week (all seizure types except for absences or myoclonias), age ≥ 6 years and no signs of self-harm. Each case will be matched to two historical controls (age +/- 5 years) from the EEG databases of the participating centres. Only those controls with two or more recorded seizures will be matched to the cases.

Intervention:

Not applicable

Main study parameters/endpoints:

Ictal asystole Ictal bradycardia Ictal QT-shortening/lengthening

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Participation does not carry risks. The sensor is wearable and miniaturised, thus minimising discomfort. If this nevertheless may occur, the study can be terminated. This study provides specific tools to investigate the seizure-related heart rate response. Subjects may thus benefit from participation by identification of otherwise unknown arrhythmias. The rationale of the study (the high SUDEP risk and the evidence in animal studies for arrhythmic cause of sudden death) specifically applies to DS, a rare epileptic syndrome including minors and incapacitated persons. The investigators believe that the lack of risks, the potential diagnostic benefit, the minimal intervention with novel and wearable sensors and the possibility to terminate the study in case of discomfort, justifies the study in this patient group.

ELIGIBILITY:
Criteria:

Cases must meet all of the following criteria:

1. DS with a known pathogenic SCN1A mutation
2. seizure frequency ≥ 1/week (all seizure types expect for absences or myoclonias)
3. no self-harm
4. age ≥ 6 years

Each case will be matched to two historical controls (age +/- 5 years). Controls will meet the following criteria:

1. definite diagnosis of epilepsy
2. no clinical suspicion of DS
3. at least two seizures recorded (all seizure types expect for absences or myoclonias) during video-EEG registration.
4. age ≥ 6 years

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the Netherlands (coordinating centre: SEIN). Procedure: The UMCU Medical Genetics department is the key referral centre in the Netherlands for DS (Brilstra, UMCU). Cases will be recruited from the UMCU database. Prior to inclusion, a panel (Gunning, Brilstra, Thijs) will review clinical data to ensure diagnostic consistency.
  Additional DS subjects will be recruited from the local DS databases at Universität Bonn (25 subjects; 4 adults; local coordinator R Surges) and UCL (100 subjects; 15 adults; local coordinator S Sisodiya).
  We will select historical controls (subjects with epilepsy without DS) from the video-EEG databases of the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Ictal asystole (sinus arrest ≥ 3 s) or ictal bradycardia (< 2nd heart rate percentile for age) | We will record heart rate patterns during seizures with miniaturized wearable EKG-monitors for 2 periods of 10 days

SECONDARY OUTCOMES:
Ictal QT lengthening or shortening | We will record heart rate patterns during seizures with miniaturized wearable EKG-monitors for 2 periods of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Roland Thijs, Dr., Principal Investigator — Stichting Epilepsie Instellingen Nederland (S.E.I.N.)
Locations (3):
- Universität Bonn, Bonn, North Rhine-Westphalia, Germany
- Stichting Epilepsie Instellingen Nederland (SEIN), Heemstede, Achterweg 5, Netherlands
- Great Ormond Street Hospital, London, South East, United Kingdom